CLINICAL TRIAL: NCT00805298
Title: Assessment of the Operative Course in Connection With Removal of Lower Third Molars With Particular Consideration to the Occurence of Pain and Swelling
Brief Title: Assessment of the Operative Course in Connection With Removal of Lower Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Tandlaegeforeningen, Calcin fonden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2008-000866-22; 01.01.08Jen
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Postoperative Pain; Inflammation
Keywords: third molar; postoperative pain; thermography; postoperative inflammation; methylprednisolone; local anaesthetic; postoperative pain after removal of lower third molars; inflammation after removal of lower third molars
MeSH Terms: conditions — Pain, Postoperative; Inflammation | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- methylprednisolone (Active Comparator)
  Interventions: Drug: methylprednisolone
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- lidocaine (Active Comparator)
  Interventions: Drug: xyloplyin adrenalin
- bupivacaine (Active Comparator)
  Interventions: Drug: marcain adrenalin

INTERVENTIONS:
Drug: methylprednisolone — 32 mg before surgery, 16 mg twice daily the day after surgery
  Other Names: medrol
  Arms: methylprednisolone
Drug: placebo — two tablets before surgery, one tablet twice daily on the day after surgery
  Arms: placebo
Drug: xyloplyin adrenalin — lidocaine local anaesthetic lidocaine 20 mg/ml, adrenalin 12,5 µg/ml maximum dosage 10 ml.
  Arms: lidocaine
Drug: marcain adrenalin — bupivacaine local anaesthetic bupivacaine 5 mg /ml, adrenaline 5 µg/ml maximum dosage 10 ml
  Arms: bupivacaine

SUMMARY:
The aim of this study is to compare postoperative complications after removal of lower third molars using two different types of anaesthetics and two different treatments against swelling and inflammation (methylprednisolone and placebo). The hypothesis is that a combination of a long-duration anaesthetic combined methylprednisolone will result in significantly less postoperative pain and inflammation.

Patients will have both lower third molars removed on two separate occasions. Each patient is randomly assigned to receive one type of local anaesthetic the first time and the other type the second time. Furthermore patients are randomised to receive either methylprednisolone or placebo the first time and the opposite treatment the second time.

During the week after surgery patients fill out a questionnaire with questions about level of pain and swelling at different times as well as the patients' perception of other postoperative complications. The patient is examined by a dentist on the 2nd and 7th day after surgery, where postoperative complications are recorded and thermographic images of the patient's face are taken to assess the degree of inflammation.

DETAILED DESCRIPTION:
Background: After removal of lower third molars complications can occur, including pain, swelling, infection and sensory disturbances. As pain intensity has been shown to be worst during the first 4-8 hours post surgery, it might be relevant to use a local anaesthetic with long duration, e.g. bupivacaine, instead of the traditionally used lidocaine. Several studies have focussed on the effect of non-steroid anti-inflammatory drugs (such as glucocorticoids, e.g. methylprednisolone) to reduce postoperative swelling. However, no studies comparing the effect of bupivacaine combined with methylprednisolone and lidocaine combined with methylprednisolone have been conducted.

Aim: To compare postoperative complications after removal of lower third molars using 1) lidocaine, 2) lidocaine combined with methylprednisolone, 3) bupivacaine and 4) bupivacaine combined with methylprednisolone.

Methods: The study compares type end extension of postoperative complications after removal of lower third molars using four different combinations of local anaesthetics and anti-inflammatory treatment. The study is conducted as a double blinded, split mouth crossover trial, where each patient has both lower third molars removed at two different occasions.

Patients are randomised to receive one type of local anaesthetic the first time and the other type the second time. Furthermore patients are randomised to receive either methylprednisolone or placebo the first time and the opposite treatment the second time.

An objective assessment of postoperative swelling and inflammation is made by means of thermographic imaging of the operated side compared to the opposite side after the operation and at 2 and 7 days post surgery.

Each patient fills out a questionnaire, where the patients' perception of pain, swelling and other complications is registered. Furthermore, complications are recorded objectively by a dentist at the 2- and 7-day post-surgery visits

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* two impacted or semi-impacted lower third molars with indication for removal
* signed informed consent

Exclusion Criteria:

* allergy to study drugs or ingredients
* need for sedation
* pregnancy
* systemic disease besides asthma/hay fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
postoperative pain | within the first week after surgery
postoperative inflammation | within the first week after surgery

SECONDARY OUTCOMES:
use of analgesics | within one week after surgery
absence from work | within one week after surgery
trismus | within one week after surgery
alveolitis (dry socket) | within one week after surgery
sensory disturbance | within one week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Christensen, DDS, Principal Investigator — University of Aarhus
Locations (1):
- School of Dentistry, Aarhus University, Aarhus, Denmark

REFERENCES:
- [Background] Beirne OR, Hollander B. The effect of methylprednisolone on pain, trismus, and swelling after removal of third molars. Oral Surg Oral Med Oral Pathol. 1986 Feb;61(2):134-8. doi: 10.1016/0030-4220(86)90173-8. PMID 3457335
- [Background] Bouloux GF, Punnia-Moorthy A. Bupivacaine versus lidocaine for third molar surgery: a double-blind, randomized, crossover study. J Oral Maxillofac Surg. 1999 May;57(5):510-4; discussion 515. doi: 10.1016/s0278-2391(99)90063-0. PMID 10319823
- [Background] Bruce RA, Frederickson GC, Small GS. Age of patients and morbidity associated with mandibular third molar surgery. J Am Dent Assoc. 1980 Aug;101(2):240-5. doi: 10.14219/jada.archive.1980.0183. PMID 6931159
- [Background] Bystedt H, Nordenram A. Effect of methylprednisolone on complications after removal of impacted mandibular third molars. Swed Dent J. 1985;9(2):65-9. PMID 3859943
- [Background] Campbell WI, Kendrick RW, Ramsay-Baggs P, McCaughey W. The effect of pre-operative administration of bupivacaine compared with its postoperative use. Anaesthesia. 1997 Dec;52(12):1212-6. PMID 9485979
- [Background] Chiapasco M, De Cicco L, Marrone G. Side effects and complications associated with third molar surgery. Oral Surg Oral Med Oral Pathol. 1993 Oct;76(4):412-20. doi: 10.1016/0030-4220(93)90005-o. PMID 8233418
- [Background] de Boer MP, Raghoebar GM, Stegenga B, Schoen PJ, Boering G. Complications after mandibular third molar extraction. Quintessence Int. 1995 Nov;26(11):779-84. PMID 8628837
- [Background] Esen E, Tasar F, Akhan O. Determination of the anti-inflammatory effects of methylprednisolone on the sequelae of third molar surgery. J Oral Maxillofac Surg. 1999 Oct;57(10):1201-6; discussion 1206-8. doi: 10.1016/s0278-2391(99)90486-x. PMID 10513866
- [Background] Holland CS. The influence of methylprednisolone on post-operative swelling following oral surgery. Br J Oral Maxillofac Surg. 1987 Aug;25(4):293-9. doi: 10.1016/0266-4356(87)90068-4. PMID 3304412
- [Background] Leone M, Richard O, Antonini F, Rousseau S, Chabaane W, Guyot L, Martin C. Comparison of methylprednisolone and ketoprofen after multiple third molar extraction: a randomized controlled study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Jan;103(1):e7-9. doi: 10.1016/j.tripleo.2006.07.005. Epub 2006 Oct 6. PMID 17178485
- [Background] Markovic AB, Todorovic L. Postoperative analgesia after lower third molar surgery: contribution of the use of long-acting local anesthetics, low-power laser, and diclofenac. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Nov;102(5):e4-8. doi: 10.1016/j.tripleo.2006.02.024. Epub 2006 Aug 10. PMID 17052624
- [Background] Mellor DJ, Mellor AH, McAteer EM. Local anaesthetic infiltration for surgical exodontia of third molar teeth: a double-blind study comparing bupivacaine infiltration with i.v. ketorolac. Br J Anaesth. 1998 Oct;81(4):511-4. doi: 10.1093/bja/81.4.511. PMID 9924222
- [Background] Mettes TG, Nienhuijs ME, van der Sanden WJ, Verdonschot EH, Plasschaert AJ. Interventions for treating asymptomatic impacted wisdom teeth in adolescents and adults. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003879. doi: 10.1002/14651858.CD003879.pub2. PMID 15846686
- [Background] Mico-Llorens JM, Satorres-Nieto M, Gargallo-Albiol J, Arnabat-Dominguez J, Berini-Aytes L, Gay-Escoda C. Efficacy of methylprednisolone in controlling complications after impacted lower third molar surgical extraction. Eur J Clin Pharmacol. 2006 Sep;62(9):693-8. doi: 10.1007/s00228-006-0164-5. Epub 2006 Aug 11. PMID 16902792
- [Background] Moore PA. Bupivacaine: a long-lasting local anesthetic for dentistry. Oral Surg Oral Med Oral Pathol. 1984 Oct;58(4):369-74. doi: 10.1016/0030-4220(84)90325-6. PMID 6387571
- [Background] Nayyar MS, Yates C. Bupivacaine as pre-emptive analgesia in third molar surgery: Randomised controlled trial. Br J Oral Maxillofac Surg. 2006 Dec;44(6):501-3. doi: 10.1016/j.bjoms.2005.09.012. Epub 2006 Feb 2. PMID 16457912
- [Background] Neal JA, Welch TB, Halliday RW. Analysis of the analgesic efficacy and cost-effective use of long-acting local anesthetics in outpatient third molar surgery. Oral Surg Oral Med Oral Pathol. 1993 Mar;75(3):283-5. doi: 10.1016/0030-4220(93)90136-r. PMID 8469535
- [Background] Osborn TP, Frederickson G Jr, Small IA, Torgerson TS. A prospective study of complications related to mandibular third molar surgery. J Oral Maxillofac Surg. 1985 Oct;43(10):767-9. doi: 10.1016/0278-2391(85)90331-3. PMID 2995624
- [Background] Renton T, Hankins M, Sproate C, McGurk M. A randomised controlled clinical trial to compare the incidence of injury to the inferior alveolar nerve as a result of coronectomy and removal of mandibular third molars. Br J Oral Maxillofac Surg. 2005 Feb;43(1):7-12. doi: 10.1016/j.bjoms.2004.09.002. PMID 15620767
- [Background] Schultze-Mosgau S, Schmelzeisen R, Frolich JC, Schmele H. Use of ibuprofen and methylprednisolone for the prevention of pain and swelling after removal of impacted third molars. J Oral Maxillofac Surg. 1995 Jan;53(1):2-7; discussion 7-8. doi: 10.1016/0278-2391(95)90486-7. PMID 7799116
- [Background] Sisk AL, Hammer WB, Shelton DW, Joy ED Jr. Complications following removal of impacted third molars: the role of the experience of the surgeon. J Oral Maxillofac Surg. 1986 Nov;44(11):855-9. doi: 10.1016/0278-2391(86)90221-1. PMID 3464711
- [Background] Skjelbred P, Lokken P. Effects of naloxone on post-operative pain and steroid-induced analgesia. Br J Clin Pharmacol. 1983 Feb;15(2):221-6. doi: 10.1111/j.1365-2125.1983.tb01489.x. PMID 6849755
- [Background] Song F, O'Meara S, Wilson P, Golder S, Kleijnen J. The effectiveness and cost-effectiveness of prophylactic removal of wisdom teeth. Health Technol Assess. 2000;4(15):1-55. PMID 10932022
- [Background] UStun Y, Erdogan O, Esen E, Karsli ED. Comparison of the effects of 2 doses of methylprednisolone on pain, swelling, and trismus after third molar surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Nov;96(5):535-9. doi: 10.1016/S1079210403004645. PMID 14600686